CLINICAL TRIAL: NCT04245215
Title: Loss of RESponse to Ustekinumab Treated by Dose Escalation
Acronym: REScUE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Belgian Inflammatory Bowel Disease Research and Development (BIRD) VZW (Other)
Collaborators: Janssen Cilag N.V./S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIRD2018001
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Crohn Disease
Keywords: dose escalation; ustekinumab
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1. Subcutaneous ustekinumab every 8 weeks (Placebo Comparator): re-induction (≈6mg/kg) intravenous ustekinumab followed by 90 mg Subcutaneous ustekinumab every 8 weeks (Q8W) for 48 weeks - receiving Q8W placebo to mimic Q4W injections
  Interventions: Drug: Ustekinumab
- 2. Subcutaneous ustekinumab every 4 weeks (Active Comparator): re-induction (≈6mg/kg) intravenous ustekinumab followed by 90 mg Subcutaneous ustekinumab every 4 weeks (Q4W) for 48 weeks
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — re-induction and dose escalation form every 8 weeks to every 4 weeks only in arm 2
  Other Names: dose escalation only in arm 2

SUMMARY:
The aim of the study is to investigate the effect of re-induction with ustekinumab ≈6mg/kg IV followed by two different maintenance dosing regimens 90 mg subcutaneous every 8 weeks (Q8W) vs 90 mg subcutaneous every 4 weeks(Q4W) on clinical, biological and pharmacological outcomes in patients with Crohn's disease who show a secondary loss of response over time

DETAILED DESCRIPTION:
The study is a prospective double blind interventional study in patients with Crohn Disease treated with ustekinumab that show an objective secondary loss of response to ustekinumab after induction treatment (>Week 16). Patients can be screened during a four week period. The screening includes a clinical, biochemical and endoscopic assessment. Patients will be randomized 8 weeks after the last subcutaneous injection with ustekinumab. All patient will receive an intravenous re-induction with ustekinumab ≈6mg/kg at baseline (8 weeks after last subcutaneous administration). After the intravenous re-induction, the patients receive either ustekinumab 90 mg subcutaneous Q4W or Q8W (altered with q8w placebo to mimic Q4W injections) till week 48. Clinical and biochemical evaluation will be planned every 8 weeks until week36 with a final evaluation at week48. Primary endpoint will be assessed at week 48. Final assessment at week 48 will include clinical, biochemical and endoscopic evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years
2. Diagnosis of Crohn's disease by endoscopic and/or radiologic examination.
3. Patient currently treated with ustekinumab, independent of previous biological exposure.
4. Patients treated with maintenance dose of ustekinumab subcutaneous 90 mg every 8 weeks
5. Documented primary response at any time point after induction (week 16) and during maintenance defined as a clinical response (physician discretion) AND confirmed by either any of the following:

   a. if biomarker elevated at start of ustekinumab (C-reactive protein>5 mg/l or fecal calprotectin >250µg/g): i. decrease of C-reactive protein by 50 % or more compared to baseline( prior to ustekinumab induction) ii. C-reactive protein <5 mg/l iii. decrease of fecal calprotectin by 50 % or more compared to baseline( prior to ustekinumab induction) iv. fecal calprotectin<250µg/g b. Documented mucosal healing (simple endoscopic score for Crohn's disease (SES-CD)<3)
6. Documented loss of response after induction (> week 16) assessed by the physician as Moderate to severe active Crohn's disease, defined as Patient Reported Outcome-2 (Abdominal Pain > 1 AND Stool Frequency > 3) AND C-reactive protein and/or fecal calprotectin increased by 25 % or more compared to the lowest value under ustekinumab treatment (C-reactive protein>5 mg/L and/or fecal calprotectin>250µg/g).
7. Presence of mucosal ulcers in at least one segment of the ileum or colon and a simple endoscopic score for Crohn's disease (SES-CD) ≥6 (for patients with isolated ileitis ≥4), as assessed by ileocolonoscopy
8. Adequate contraception in female of reproductive age
9. Have the capacity to understand and sign an informed consent form.
10. Be able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Ongoing treatment with

   1. other concomitant biological (vedolizumab, anti-TNF)
   2. Steroids >20 mg prednisolone or equivalent at baseline (budesonide >6 mg)
   3. Patient already receiving ustekinumab every 4 weeks
2. Women that are pregnant, nursing, or planning pregnancy
3. Have screening laboratory test results within the following parameters:

   1. Haemoglobin < 8.5 g/dL
   2. Platelets < 100,000 /mm3
   3. Serum creatinine ≥ 1.7 mg/dL
   4. aspartate aminotransferase and alanine aminotransferase > 3 times the upper limit of normal range
   5. Direct (conjugated) bilirubin ≥ 3.0 mg/dL.
4. Have current signs or symptoms of infection confirmed by positive stool or blood testing (including gastrointestinal pathogens, tuberculosis, human immunodeficiency virus, hepatitis B, hepatitis C).
5. Patients with a positive stool sample for gastrointestinal pathogen including Clostridium difficile.
6. Evidence of current or previous clinically significant disease, medical condition other than Crohn's Disease, finding of the medical examination, or laboratory value at the screening visit outside the reference range that is of clinical relevance, that in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data.
7. Patients with an ileostomy
8. Patients that received an intravenous re-induction with ustekinumab within the 6 months prior to baseline.
9. Patients with an impassable stenosis even after attempt of endoscopic balloon dilation.
10. Patients with an abscess

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with steroid free clinical remission and fecal calprotectin<250µg/g at week 48 | week 48
  Proportion of patients with steroid free clinical remission (patient reported outcome-2 remission: abdominal pain ≤ 1 AND stool frequency ≤ 3) and fecal calprotectin<250µg/g at week 48. [stool frequency (ST): average number of liquid stools for 1 week abdominal pain (AP): average scoring for abdominal pain for 1 week (0=none; 1=mild, 2=moderate; 3= severe)]

SECONDARY OUTCOMES:
Proportion of patients with complete endoscopic remission at week 48 | week 48
  Proportion of patients with complete endoscopic remission (simple endoscopic score for Crohn's disease (SES-CD )<3) at week 48
Proportion of patients with endoscopic remission at week 48 | week 48
  Proportion of patients with endoscopic remission (simple endoscopic score for Crohn's disease (SES-CD) <5) at week 48
Proportion of patients with endoscopic response at week 48 | week 48
  Proportion of patients with endoscopic response (≥50% decrease in simple endoscopic score for Crohn's disease (SES-CD)) at week 48
Proportion of patients with clinical remission at week 48 | week 48
  Proportion of patients with clinical remission (patient reported outcome-2 remission: abdominal pain ≤ 1 AND stool frequency ≤ 3) at week 48
Proportion of patients with biomarker remission at week 48 | week 48
  Proportion of patients with biomarker remission (C-reactive protein <5 mg/L and fecal calprotectin <250 µg/g) at week 48
Proportion of patients with at all time points after baseline ustekinumab trough concentration > 1.4 μg/mL | between baseline and week 48
  Proportion of patients with at all time points after baseline ustekinumab trough concentration > 1.4 μg/mL
Proportion of patients with serious adverse events at week 48 | Week 48
  Proportion of patients with serious adverse events at week 48

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bossuyt, MD, Principal Investigator — BIRD (Belgian IBD Research and Development) vzw
Locations (1):
- Ingrid Arijs, Zaventem, Belgium

IPD SHARING:
Plan to Share IPD: No